CLINICAL TRIAL: NCT03578276
Title: Lessdrops™ Prophylactic Treatment After Routine Phacoemulsification Compared to Standard Drops Regimen
Brief Title: Prophylactic Treatment: Lessdrops™ vs Standard Drops Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carolina Eyecare Physicians, LLC (Other)
Collaborators: Science in Vision (Other); Imprimis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEP 2016-001
Record Dates: First submitted 2018-06-19; First posted 2018-07-06 (Actual); Results first posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Cataract
Keywords: cataract surgery; Prophylaxis
MeSH Terms: conditions — Cataract | interventions — prednisolone acetate; bromfenac

STUDY DESIGN:
Intervention Model Description: Participants' eyes are assigned to one of two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LessDrops (Active Comparator): Compounded eye drop containing Gatifloxacin (antibiotic), bromfenac (non-steroidal anti-inflammatory), and prednisolone acetate 1% used three times a day (TID) starting 1 day prior to surgery and continuing after surgery for 2 weeks then twice a day for a week and once a day for another week.
  Interventions: Drug: Pred-Gati-Brom
- Standard of Care (Active Comparator): * Gatifloxacin 0.5%, 1 drop, QID for 3 days prior to surgery and will continue for 2 weeks after surgery and then discontinue.
  * Bromfenac 0.07%: 1 drop QD starting 3 days before surgery, continue QD for 4 weeks after surgery and then discontinue.
  * Prednisolone acetate 1% will be started after surgery QID for 2 weeks, tapered to BID for 2 weeks, and then discontinue.
  Interventions: Drug: Prednisolone acetate 1% ophthalmic suspension; Drug: Gatifloxacin Ophthalmic; Drug: Bromfenac 0.075% Oph Solution

INTERVENTIONS:
Drug: Pred-Gati-Brom — The combination drop therapy containing prednisolone acetate 1%, gatifloxacin 0.5%, and bromfenac 0.075%
  Other Names: LessDrops
  Arms: LessDrops
Drug: Prednisolone acetate 1% ophthalmic suspension — Steroidal anti-inflammatory
  Arms: Standard of Care
Drug: Gatifloxacin Ophthalmic — Antibiotic
  Arms: Standard of Care
Drug: Bromfenac 0.075% Oph Solution — Non-steroidal anti-inflammatory
  Arms: Standard of Care

SUMMARY:
To compare the use of a compounded eye drop containing an antibiotic, a non-steroidal and steroidal anti-inflammatory to standard of care that is the use of 3 different topical medications to prevent inflammation and infection after routine cataract surgery.

DETAILED DESCRIPTION:
Cataract surgery is one of the most commonly performed surgeries in the world today. To improve the overall procedure outcome, prophylactic topical antibiotics and anti-inflammatories (steroidal and non-steroidal, NSAID) are frequently used to decrease the risk of postoperative infection (e.g., endophthalmitis) and intraocular inflammation (e.g., macular edema, CME).

Even though, the large body of literature that supports the significance of prophylactic eye drops prior to surgery, patient compliance is a common problem. Different factors have been associated with patient's lack of compliance. It could be due to patient's inability to self- administer the drops, lack of understanding of the importance of using the prophylactic treatment as well as understanding the instructions of how to administer the drops and its storage, or just forgetfulness or the fact that they don't like to put the drops multiple times a day for 2-4 weeks, therefore they just avoid doing it. About 64% of patients adhere to the prescribed treatment.

There is a new alternative that combines the most commonly used antibiotic and anti-inflammatories into a single drop. The use of a single drop compounded ophthalmic solution may offer advantages such as increased compliance, patient comfort and reduced ocular toxicity. T

The purpose of this study is to compare the Pred-Gati-Brom formulation to the standard topical drops regimen that includes the topical use of Gatifloxacin, Bromfenac and Prednisolone acetate 1%.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing bilateral cataract extraction or refractive lens exchange with intraocular lens implantation.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Willing and able to administer eye drops and record the times the drops were instilled.
* Scheduled to undergo standard cataract surgery with topical anesthesia in both eyes within 6-15 days between surgeries.
* Potential postoperative best-corrected visual acuity of 20/30 or better.

Exclusion Criteria:

* Severe preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmos or macrophthalmos, optic nerve atrophy, advanced macular degeneration, advanced glaucomatous damage, etc.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/noninfectious conjunctivitis, keratitis or uveitis.
* History of chronic intraocular inflammation.
* History of retinal detachment.
* Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
* Any additional ocular surgical procedures at time of cataract extraction (i.e. iStent) except corneal incisions for the correction of astigmatism.
* Anesthesia other than topical anesthesia (i.e. retrobulbar, general, etc).
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
* Participation in (or current participation) any ophthalmic investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Solomon, MD, Principal Investigator — Carolina Eyecare Physicians, LLC
Locations (1):
- Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Standard of Care: * Gatifoxacin 0.5%, 1 drop, QID for 3 days prior to surgery and will continue for 2 weeks after surgery and then discontinue.
  * Bromfenac 0.07%: 1 drop QD starting 3 days before surgery, continue QD for 4 weeks after surgery and then discontinue.
  * Prednisolone acetate 1% will be started after surgery QID for 2 weeks, tapered to BID for 2 weeks, and then discontinue.
  Prednisolone acetate 1% ophthalmic suspension: Steroidal anti-inflammatory
  Gatifloxacin Ophthalmic: Antibiotic
  Bromfenac 0.075% Oph Solution: Non-steroidal anti-inflammatory
Period: Overall Study
Arm/Group | LessDrops | Standard of Care
Started | 35; 35 Eyes | 35; 35 Eyes
Completed | 33; 33 Eyes | 33; 33 Eyes
Not Completed | 2; 2 Eyes | 2; 2 Eyes
Not completed — Subjects did not comply with study protocol instructions. | 2 | 2

BASELINE CHARACTERISTICS:
Population: 33 subjects were enrolled, with 66 eyes. Subjects had one eye in each of the two arms.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | LessDrops | Standard of Care | Total
Number analyzed (Participants) | 33 | 33 | 33
Number analyzed (Eyes) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (6.6) | 69.7 (6.6) | 69.7 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 33 | 33 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 35 subjects signed the informed consent and who met the inclusion/exclusion criteria were successfully enrolled in the study.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 5 | 5 | 10
    White | 28 | 28 | 56
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Preoperative Exam) in Macular Thickness
Description: Thickness of the macula measured in microns, recorded as the change from baseline.
Time Frame: Month 1
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: eyes
Arm/Group | LessDrops | Standard of Care
Number analyzed (Participants) | 33 | 33
Number analyzed (eyes) | 33 | 33
microns | 4.91 (8.46) | 1.30 (4.13)

2. Secondary Outcome: Change From Baseline (Preoperative Exam) in Pachymetry (Corneal Thickness)
Description: Thickness of the cornea measured in microns, measured as the change from baseline
Time Frame: Month 1
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | LessDrops | Standard of Care
Number analyzed (Participants) | 33 | 33
Number analyzed (Eyes) | 33 | 33
microns | 3.18 (20.46) | 0.63 (18.37)

3. Secondary Outcome: Change From Baseline (Preoperative Exam) in Intraocular Pressure (IOP)
Description: Measurement of the pressure inside the eye in mmHg, recorded as the change from baseline
Time Frame: Month 1
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | LessDrops | Standard of Care
Number analyzed (Participants) | 33 | 33
Number analyzed (eyes) | 33 | 33
mmHg | -0.33 (3.35) | -0.21 (3.37)

ADVERSE EVENTS:
Time Frame: One month
Arm/Group | LessDrops | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 2/33 | 6/33
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LessDrops (N=33) | Standard of Care (N=33)
High intraocular pressure (Eye disorders) | 1 | 2
Rebound inflammation (Eye disorders) | 1 | 2
Macular edema (Eye disorders) | 0 | 1
Punctate epithelial erosions (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT03578276/Prot_SAP_000.pdf